CLINICAL TRIAL: NCT05158959
Title: Study of the Association Between Renal Reserve Function and Progression of Renal Function to Predict Chronic Kidney Disease Risk in Thai Elderly
Brief Title: Association Between Renal Reserve Function and Progression of Renal Function to Predict CKD Risk in Thai Elderly
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Kearkiat Praditpornsilpa, Professor of Medicine, Chulalongkorn University
Other Study IDs: IRB NO.527/62
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-09

CONDITIONS: Elder; Renal Function Abnormal
Keywords: Renal functional reserve, CKD progression, Elderly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study investigates renal functional reserve in elderly.

DETAILED DESCRIPTION:
The prevalence of CKD in elder is high as age has been a variable in eGFR equation. eGFR by calculation always declines in parallel with age. The assumption that a persistent over 3 months of eGFR less than 60 mL/min/1.73m2 define CKD with risk of progression and need refer to nephrologist may not necessary true in aging population. We study renal functional reserve in elderly population who risk of CKD progression and ESRD is the highest prevalence in human life cycle and explore whether renal functional reserve can be used as ad additional marker of CKD progression in elderly.

ELIGIBILITY:
Inclusion Criteria:

* Patient age > 60 years at screening
* Patient willing to participate in the study and can provide inform consent
* Patient have residual kidney function ≤ 90 ml/min/1.73m2 by CKD-EPI equation

Exclusion Criteria:

* Patient active smoking
* Patient have Charlson comorbidity index > .....
* Patient active cancer
* Patient contraindications for blood collection
* Patients with a history of hypersensitivity to cimetidine or amino acid IV solution

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elders age more than 60 years who are non-frail and has no limited life expectancy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-10-24 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of renal functional reserve per 12 months (mL/min) | 12 months
  Renal functional reserve defined as the difference between baseline creatinine clearance and creatinine clearance achieved under stimulation with amino acid infusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Kearkiat Praditpornsilpa, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No